CLINICAL TRIAL: NCT03350607
Title: Observational Prospective Monocentric Study Evaluating "Sweeper" Use During Epiretinal Membrane Surgery
Brief Title: " Sweeper " and Epiretinal Membrane Surgery
Acronym: SWEEPING
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0295
Record Dates: First submitted 2017-11-14; First posted 2017-11-22 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Epiretinal Membrane
Keywords: Epiretinal membrane, sweeper, forceps, microperimetry
MeSH Terms: conditions — Epiretinal Membrane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non interventional study — Non interventional study (collect of data)

SUMMARY:
Epiretinal membrane (ERM) is a pathological phenomenon requiring surgery when vision is altered.

ERM surgery requires ERM peeling, then active internal limiting membrane (ILM) peeling if it is not spontaneously peeled with ERM. Initiation of peeling is very delicate and can lead to micro scotoma when realized with microscopic forceps. The Sweeper is a microscopic tool with a soft silicon tip covered with diamond dust which allows peeling initiation without retina prehension. It may reduce retinal trauma and visual sequelae.

Purpose of our study is to evaluate use of sweeper during 20 ERM surgeries. The investigator will compare microperimetry before surgery versus those after 1 month (M1) and 3 months (M3), and measure difference of number and depths of micro scotoma.

The investigator will note: number of forceps uses if sweeper is inefficient and all areas of sweeper use to correlate them with micro scotoma.

The investigator will evaluate visual and optical coherence tomography improvement after surgery.

DETAILED DESCRIPTION:
Epiretinal membrane (ERM) is a pathological phenomenon that leads to visual loss, visual distortions, central scotoma, and diplopia. No medical treatment is yet available.

ERM surgery requires separation of normal retina and epiretinal membrane. After epiretinal peeling, if internal limiting membrane (ILM) is not spontaneously peeled with ERM, surgeon peels ILM from retina (also named active peeling). Initiation of peeling is very accurate and delicate. Either microscopic forceps or sweeper are used to initiate peeling. Sweeper is a microscopic tool with a soft silicon tip covered with diamond dust which allows peeling initiation without retina prehension. It may reduce retinal trauma and visual sequelae.

ILM active peeling reduces recurrence of ERM and rate of repeat surgery. No visual acuity loss has been found. But 2 studies show increase of micro scotoma at micro-perimetry after active ILM peeling with forceps.

Purpose of our study is to evaluate use of sweeper during 20 ERM surgeries. The investigator will compare microperimetry before surgery versus those after 1 month (M1) and 3 months (M3), and measure difference of number and depths of micro scotoma.

The investigator will note: number of forceps uses if sweeper is inefficient, all areas of sweeper use to correlate them with micro scotoma.

The investigator will evaluate visual and optical coherence tomography improvement after surgery.

Our study doesn't include any intervention while surgeries would be realized with or without study participation. Examinations are non-invasive, usual, and done during usual medical visit without additional visit.

ELIGIBILITY:
Inclusion Criteria:

* consent,
* adult patient,
* Epiretinal membrane

Exclusion Criteria:

* perimetry impossible

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The population concerned corresponds to the major patients consulting in the ophthalmology department at the Nantes University Hospital and presenting an epiretinal membrane and an operative indication.
  Patients will be included at the epiretinal membrane surgery programming consultation. No inclusion will be made as part of the emergency.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2018-01-24 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Difference of number and depth of micro scotoma before and after epiretinal membrane (ERM) surgery with sweeper | microperimetry at baseline, then 1 month after surgery (M1), then 3 months after (M3)

SECONDARY OUTCOMES:
Efficacy of sweeper mesured by number of forceps uses if sweeper is inefficient | Day of surgery
Visual improvement measured by visual acuity and optical coherence tomography improvement after surgery , visual acuity and OCT morphometry before surgery, M1 and M3 | at baseline, then 1 month after surgery (M1), then 3 months after (M3)
Optical coherence tomography (OCT) improvement after surgery measured by OCT morphometry | at baseline, then 1 month after surgery (M1), then 3 months after (M3)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Baptiste Ducloyer, Dr, Principal Investigator — Nantes University Hospital
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

REFERENCES:
- [Background] Azuma K, Ueta T, Eguchi S, Aihara M. EFFECTS OF INTERNAL LIMITING MEMBRANE PEELING COMBINED WITH REMOVAL OF IDIOPATHIC EPIRETINAL MEMBRANE: A Systematic Review of Literature and Meta-Analysis. Retina. 2017 Oct;37(10):1813-1819. doi: 10.1097/IAE.0000000000001537. PMID 28207608
- [Background] Fang XL, Tong Y, Zhou YL, Zhao PQ, Wang ZY. Internal limiting membrane peeling or not: a systematic review and meta-analysis of idiopathic macular pucker surgery. Br J Ophthalmol. 2017 Nov;101(11):1535-1541. doi: 10.1136/bjophthalmol-2016-309768. Epub 2017 Mar 17. PMID 28314834
- [Background] Ripandelli G, Scarinci F, Piaggi P, Guidi G, Pileri M, Cupo G, Sartini MS, Parisi V, Baldanzellu S, Giusti C, Nardi M, Stirpe M, Lazzeri S. Macular pucker: to peel or not to peel the internal limiting membrane? A microperimetric response. Retina. 2015 Mar;35(3):498-507. doi: 10.1097/IAE.0000000000000330. PMID 25158943
- [Background] Deltour JB, Grimbert P, Masse H, Lebreton O, Weber M. DETRIMENTAL EFFECTS OF ACTIVE INTERNAL LIMITING MEMBRANE PEELING DURING EPIRETINAL MEMBRANE SURGERY: Microperimetric Analysis. Retina. 2017 Mar;37(3):544-552. doi: 10.1097/IAE.0000000000001179. PMID 27429376